CLINICAL TRIAL: NCT03565874
Title: Heart Rate Variability Biofeedback (HRVB) With Mothers Who Delivered a Preterm Infant: A Feasibility Study
Brief Title: Heart Rate Variability and Prematurity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Urben Sébastien, Head of Research Unit, University Service of Child and Adolescent Psychiatry, University of Lausanne Hospitals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2017-02199
Record Dates: First submitted 2018-03-20; First posted 2018-06-21 (Actual); Results first posted 2019-08-29 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Premature Birth; Maternal Distress - Delivered; Stress; Anxiety
MeSH Terms: conditions — Premature Birth; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heart Rate Variability Biofeedback (Experimental): HRVB program conducted over the course of 2 weeks of individual daily exercises for 20 minutes per day.
  Interventions: Device: Heart rate variability biofeedback

INTERVENTIONS:
Device: Heart rate variability biofeedback — Before the start of the program and after one week of adherence to the program, two sessions will be conducted with a psychologist in order to define each participant's individual resonance frequency (i.e., breathing rhythm allowing for cardiac coherence), using the Nexus program from Mindmedia company. Then, each participant will receive training on the HRVB program using an Emwave device. The HRVB program itself will be carried individually for 20 min daily over the course of two weeks. Five daily sessions of 10 minutes will be considered as the minimum adherence to the program. Each participant will be asked to report in a diary all eventual major stressful life events.

SUMMARY:
Mothers who deliver prematurely (<37 weeks of gestational age) experience intense stress and anxiety given that their child's survival and development might be compromised. From the existing literature, it is known that a heart rate variability biofeedback (HRVB) program increases heart rate variability (HRV), which in turn, is related to significant reductions in perceived stress and anxiety. This study's aim is to evaluate the feasibility of an HRVB program in a sample of mothers who delivered prematurely.

ELIGIBILITY:
Inclusion Criteria:

* Delivery between 33 and 37 weeks of gestational age
* Living in Lausanne or surroundings
* Infant is expected to survive
* Singleton birth
* Consent of mother to participate in the study
* Sufficient French-speaking skills to fill out the questionnaires
* Mothers older than 18 years of age

Exclusion Criteria:

* Infant with cranial abnormality/neurological squeal such as cystic periventricular leukomalacia (PVL) and intraventricular haemorrhage (IVH)
* Maternal history of drug or alcohol abuse or severe psychiatric disorders before or during pregnancy
* Infant with congenital anomalies
* Infant with hearing or vision loss
* Mother and infant participating in another clinical trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Urben, PhD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitaliter Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Heart Rate Variability Biofeedback
Started | 6
Completed | 4
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Heart Rate Variability Biofeedback
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Switzerland | 6

OUTCOME MEASURES:

1. Primary Outcome: Feasibility: Acceptance (Ratio)
Description: The ratio of acceptance of study participation (number of participants who accept to participate to the study / number of participants to whom the study has been proposed) * 100
Time Frame: After completing the HRVB program (on average 3 weeks)
Population: We propose the study to 18 participants and 6 accept to participate. Ratio: (6/18)*100
Measure: Number; unit: percentage of <participants>
Arm/Group | Heart Rate Variability Biofeedback
Number analyzed (Participants) | 18
percentage of <participants> | 33.3

2. Primary Outcome: Feasibility: Drop-out
Description: The ratio of drop out.
Time Frame: After completing the HRVB program (on average 3 weeks)
Measure: Number; unit: percentage of participants
Arm/Group | Heart Rate Variability Biofeedback
Number analyzed (Participants) | 6
percentage of participants | 33.3

3. Primary Outcome: Feasibility: Number of Sessions Completed During Study
Description: Compliance with study protocol regarding the number of sessions attended by the participants.
Time Frame: After completing the HRVB program (on average 3 weeks)
Measure: Mean (Standard Deviation); unit: sessions completed
Arm/Group | Heart Rate Variability Biofeedback
Number analyzed (Participants) | 4
sessions completed | 10.25 (0.96)

4. Primary Outcome: Satisfaction Regarding the Intervention
Description: Satisfaction will be measured through a questionnaire. Questions will be asked about global satisfaction, utility, timing and difficulty about their experience (assessed on single item Likert scale).
  Higher scores reflects more satisfaction. Possible range 2 to 10.
Time Frame: After completing the HRVB program (on average 3 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Heart Rate Variability Biofeedback
Number analyzed (Participants) | 4
score on a scale | 7.5 (0.57)

5. Secondary Outcome: HRV: RMSDD
Description: The root-mean square differences of successive R-R intervals (RMSDD) will be used as measures to assess HRV level before and after participation in the HRVB program.
Time Frame: Before and after completing the HRVB program (on average 3 weeks).
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Heart Rate Variability Biofeedback
Number analyzed (Participants) | 4
milliseconds
  Before intervention | 42.7 (24.76)
  After intervention | 49.13 (37.04)

6. Secondary Outcome: HRV: HF
Description: High Frequency (HF) will be used as measures to assess HRV level before and after participation in the HRVB program.
Time Frame: Before and after completing the HRVB program (on average 3 weeks).
Measure: Mean (Standard Deviation); unit: high frequency power normalized unit
Arm/Group | Heart Rate Variability Biofeedback
Number analyzed (Participants) | 4
high frequency power normalized unit
  Before intervention | 45.63 (11.16)
  After intervention | 27.81 (14.12)

7. Secondary Outcome: Stress
Description: Perceived stress will be measured on the Perceived Stress Scale-14 (PSS-14). PSS-14 score is calculated on 14 items ranging from 0 to 4. The 7 positive state items (4,5,6,7,9,10 and 13) must have their score reversed (0=4, 1=3, 2=2, 3=1, 4=0) in order to calculate the total score by summing up all 14 items.(Min=0, Max=56). Higher scores indicate a higher level of stress. A validated French version of the PSS will be used.
Time Frame: Before and after completing the HRVB program (on average 3 weeks).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Heart Rate Variability Biofeedback
Number analyzed (Participants) | 4
score on a scale
  Before intervention | 29 (9.97)
  After intervention | 19.75 (14.24)

8. Secondary Outcome: PTSD
Description: Post-traumatic stress disorder symptoms will be measured with the Post-traumatic stress disorder checklist (PCL-5) for Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (DSM-5). PCL-5 is a 20 items self-report measure that assesses the presence and severity of PTSD symptoms. Items on the PCL-5 correspond to DSM-5 criteria for PTSD. Each item is rated on a 5 point Likert scale (from "Not at all" to "Extremely"). Total score is calculated by adding up scores for all items (Min = 0, Max = 80). Higher scores indicate a higher level of PTSD. A validated French version of the PCL will be used.
Time Frame: Before and after completing the HRVB program (on average 3 weeks).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Heart Rate Variability Biofeedback
Number analyzed (Participants) | 4
score on a scale
  Before intervention | 27.75 (15.73)
  After intervention | 16.25 (12.69)

9. Secondary Outcome: Anxiety
Description: Anxiety symptoms will be measured with the State and Trait Anxiety Inventory (STAI). STAI score is calculated on 40 items (20 items assessing trait anxiety and 20 items assessing state anxiety) rated on a 4 point Likert scale (from "Almost never" to "Almost always"). Total score for state and trait anxiety is calculated by adding up all items (Min = 20, Max = 80).
  Higher scores indicate a higher level of anxiety. A validated French version of the STAI will be used.
Time Frame: Before and after completing the HRVB program (on average 3 weeks).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Heart Rate Variability Biofeedback
Number analyzed (Participants) | 4
score on a scale
  STAI trait - Before intervention | 32.75 (8.46)
  STAI trait - After intervention | 32.25 (6.65)
  STAI state - Before intervention | 49.25 (18.46)
  STAI state - After intervention | 34.5 (7.59)

10. Secondary Outcome: Depression
Description: Depression symptoms will be assessed with a 13-item short form of the Beck Depression Inventory (BDI), which is a 13-item, self-report rating inventory that measures symptoms of depression. The scale for each item goes from 0 to 3.
  Total score is calculated by adding up scores from each item (Min = 0, Max = 39).
  Higher scores indicate a higher level of depression. A validated French version of the BDI will be used.
Time Frame: Before and after completing the HRVB program (on average 3 weeks).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Heart Rate Variability Biofeedback
Number analyzed (Participants) | 4
score on a scale
  Before intervention | 4.75 (4.57)
  After intervention | 3.5 (1)

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Heart Rate Variability Biofeedback
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/74/NCT03565874/Prot_SAP_000.pdf